CLINICAL TRIAL: NCT01069497
Title: Impact of a Multifaceted Intervention on the Preventability of Infections in Residents of French Nursing Homes: Cluster-randomised Controlled Trial (ENLIL Study)
Brief Title: Preventability of Infections in Residents of French Nursing Homes
Acronym: ENLIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Observatoire du Risque Infectieux en Gériatrie (Other)
Collaborators: Ministry of Health, France (Other Government); Pierre Fabre Laboratories (Industry); Gaba Laboratories (Other)
Responsible Party: Monique Rothan-Tondeur, Observatoire du Risque Infectieux en Gériatrie
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V15
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2009-09

CONDITIONS: Infection Control
Keywords: Infection control; Urinary Tract Infections; Respiratory Tract Infections
MeSH Terms: conditions — Urinary Tract Infections; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Nursing Homes (Experimental): Comprising 24 nursing homes implementing a specific infection prevention program
  Interventions: Other: Prevention of infections program
- Usual care Nursing Homes (No Intervention)

INTERVENTIONS:
Other: Prevention of infections program — The intervention mainly involves implementing urinary, respiratory and gastrointestinal infection prevention measures. Study nursing home medical coordinators will be in charge of training their own teams. For this, they will be provided with:
  * a slide-show of recommendations (commented by an expert),
  * recommendations guides (on paper and on computer) to be shown to their teams. Means will be provided to the intervention nursing homes : Hydro-alcoholic solutions, disinfectant detergent-impregnated tissues, mouth care kits, tec.
  Arms: Intervention Nursing Homes

SUMMARY:
STUDY HYPOTHESIS : An infection prevention program adapted for the nursing home context can reduce by 5% the number of infections (urinary, upper and lower respiratory and gastrointestinal) in elderly residents in nursing homes.

STUDY DESIGN : The proposal is for an interventional cluster (nursing home) study comprising 2 randomized groups: group 1 (interventional), comprising 25 nursing homes implementing a specific infection prevention program; and group 2 (control), 25 nursing homes continuing to implement their routine prevention measures.

ELIGIBILITY:
Inclusion Criteria:

* Nursing homes which contain a medical coordinator and at least one nurse and/or nursing auxiliary.
* Nursing Homes located in France (North-West)
* All the residents present or entering the facility during the study period

Exclusion Criteria:

* Nursing homes where a prevention program has already been implemented

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Number of infections (urinary, upper and lower respiratory and gastrointestinal) in elderly residents in nursing homes | every month

SECONDARY OUTCOMES:
Number of death | every month
Number of hospitalizations | every month
Number of of prescriptions for antimicrobials | every month

CONTACTS AND LOCATIONS:
Overall Officials: Monique Rothan Tondeur, PhD, Principal Investigator — ORIG, EHESP

REFERENCES:
- [Derived] Chami K, Gavazzi G, Bar-Hen A, Carrat F, de Wazieres B, Lejeune B, Armand N, Rainfray M, Hajjar J, Piette F, Rothan Tondeur M. A short-term, multicomponent infection control program in nursing homes: a cluster randomized controlled trial. J Am Med Dir Assoc. 2012 Jul;13(6):569.e9-17. doi: 10.1016/j.jamda.2012.04.008. Epub 2012 Jun 7. PMID 22682697